CLINICAL TRIAL: NCT03902106
Title: Physiological Response to Salbutamol and Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SALB
Record Dates: First submitted 2019-03-26; First posted 2019-04-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Healthy
MeSH Terms: interventions — Albuterol; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- beta2-agonist and exercise (Active Comparator): Subjects undergo exercise training with administration of salbutamol (800 microgram in 12 hours x 2)
  Interventions: Drug: salbutamol; Other: exercise
- placebo and exercise (Sham Comparator): Subjects undergo exercise training with administration of sham placebo
  Interventions: Other: exercise

INTERVENTIONS:
Drug: salbutamol — subjects ingest salbutamol
  Arms: beta2-agonist and exercise
Other: exercise — subjects undergo 6 weeks of endurance training (3 times weekly)

SUMMARY:
The scope of the study is to investigate the physiological response to salbutamol and exercise. A particular focus is on the metabolic response and amine metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* VO2max of >55 ml/min/kg for men and >50 ml/min/kg for women
* Body mass index (BMI) < 26

Exclusion Criteria:

* Chronic use of beta2-agonist or allergy towards beta2-agonist
* Serious adverse effects to beta2-agonist
* Chronic disease deemed by the study responsible medical doctor to interfere with any part of the study
* Smoking
* Chronic use of prescription medicine deemed by the study responsible medical doctor to interfere with any part of the study
* Pregnancy (for women)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Body composition | Baseline, 2 weeks, 4 weeks and 6 weeks
  Change in body composition (measured by dual energy x ray absorptiometry)
Maximal oxygen consumption (VO2max) | Baseline, 2 weeks, 4 weeks and 6 weeks
  Change in VO2max (measured during bike ergometer cycling to exhaustion)

SECONDARY OUTCOMES:
Salbutamol urine concentration | Before (baseline) as well as 0-1 hours, 1-2 hours, 2-4 hours, 4-8 hours, and 8-16 hours after administration
  Concentration of salbutamol in urine

OTHER OUTCOMES:
Muscle strength | Baseline, 2 weeks, 4 weeks and 6 weeks
  Isometric muscle force of the quadriceps

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No